CLINICAL TRIAL: NCT01872897
Title: A Multi-centred, Randomised, Open Label, Placebo-controlled, Two-period Crossover Study to Evaluate 4-hour Esophageal pH Change in GERD Patients After Administration of Compound Sodium Alginate Double Action Chewable Tablets or Matching Placebo Tablets
Brief Title: Compound Sodium Alginate Double Action Chewable Tablets 4-hour Esophageal pH Study in GERD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GA1202
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; GERD; Acid reflux; Compound Sodium Alginate Double Action Chewable Tablet; Gaviscon Double Action Tablets
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Alginate Double Action Chewable Tablets, then Placebo tablets (Active Comparator): 4 Compound Sodium Alginate Double Action Chewable Tablets administered as a single dose, followed by 7 days of Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily), then a single dose of 4 Placebo tablets
  Interventions: Drug: Sodium Alginate Double Action Chewable Tablets
- Placebo tablets, then Sodium Alginate Double Action Chewable Tablets (Placebo Comparator): Single dose of 4 Placebo tablets, followed by 7 days of Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily), then a single dose of 4 Compound Sodium Alginate Double Action Chewable Tablets
  Interventions: Drug: Sodium Alginate Double Action Chewable Tablets; Drug: Placebo

INTERVENTIONS:
Drug: Sodium Alginate Double Action Chewable Tablets — 4 tablets as a single dose
  Other Names: Gaviscon Double Action Tablets
Drug: Placebo — 4 tablets as a single dose
  Arms: Placebo tablets, then Sodium Alginate Double Action Chewable Tablets

SUMMARY:
This study is being conducted to assess the effectiveness of the Compound Sodium Alginate Double Action Chewable Tablets compared to placebo on acidic reflux events into the esophagus in patients diagnosed with Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* meets the diagnostic criteria for GERD with a GERD history of frequent episodes of GERD-related symptoms during the last 2 months prior to study screening. The patient must also meet the following criteria:

  1. The only or main symptom is heartburn (burning feeling back of breast bone) and/or acid reflux. Symptoms persist or have occurred repeatedly for more than 2 months;
  2. As assessed by the Investigator at screening by questioning of the patient, the frequency of occurrence of heartburn is ≥ 3 days/week and the score of severity of heartburn in general is ≥ moderate within 3 weeks before screening

Exclusion Criteria:

* Patients who have a history of drug, solvent or alcohol abuse (weekly alcohol intake ≥ 140 g).
* Patients who have suffered cardiac chest pain within the last year.
* Patients who have suffered a recent, significant unexplained weight loss of more than 6 kg in the last 6 months.
* Female patients of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Pregnancy or lactating mother.
* Patients with a history and/or symptom profile suggestive of the following: any other gastrointestinal (GI) disease, erosive GERD (Los Angeles [LA] classification grades C-D), Barrett's oesophagus, acute peptic ulcer and/or ulcer complications, Zollinger-Ellison syndrome, gastric carcinoma, pyloric stenosis, oesophageal or gastric surgery, intestinal obstruction, current pernicious anaemia, indication for H. pylori eradication therapy, known gastrointestinal bleeding (hematochezia or hematemesis) within the last 3 months, and severe diseases of other major body systems.
* Patients who are observed at screening to have a hiatus hernia with a diameter which exceeds 3 cm.
* Patients who have taken anti-cholinesterase drugs, traditional Chinese medicines for treating gastrointestinal disease, ulcerlmin or misoprostol preparations within 7 days prior to screening or throughout the study.
* Patients who have taken PPIs during the 10 days prior to screening, prokinetics or H2 antagonists during the 5 days prior to screening or systemic glucocorticosteroids, non-steroidal anti-inflammatory drugs (except for low dose aspirin which can be given for cardioprotection) on more than 3 consecutive days or PPI-based triple or quadruple therapy for eradication of H. pylori during the last 28 days.
* Patients taking or requiring to take macrolide antibiotics, such as erythromycin, azithromycin, from the day before screening.
* Patients with difficulty in swallowing.
* Patients with known hypophosphataemia, phenylketonuria or hypercalcaemia.
* Patients with severe constipation, or history of intestinal obstruction.
* In the opinion of the Investigator, patients with damaged heart or kidney function and patients who require a low sodium diet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yaozong, MD, PhD, Principal Investigator — Shanghai Jiao Tong University, School of Medicine, Shanghai, China
Locations (1):
- RB Investigational Sites, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Participants in Group A received a single dose (four tablets) of Sodium Alginate Double Action Chewable Tablets at Visit 2, followed by 7 days of Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily) and a single dose (four tablets) of Placebo tablets at Visit 3.
- Group B: Participants in Group B received a single dose (four tablets) of placebo tablets at Visit 2, followed by 7 days of Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily) and a single dose (four tablets) of Sodium Alginate Double Action Chewable Tablets at Visit 3.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 22 | 23
Completed | 21 | 23
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (15.27) | 39.3 (16.90) | 40.4 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 11 | 15 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0 | 0 | 0
  Asian | 22 | 23 | 45
  Afro-Caribbean | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time During the 4-hour Post-dosing Period With pH Below pH 4
Description: The primary efficacy endpoint will be the percentage of time during the 4-hour post-dosing period with pH below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time with pH below pH 4
Groups:
- Sodium Alginate Double Action Chewable Tablets: Results from all subjects following dosing with Sodium Alginate Double Action Chewable Tablets
- Placebo Tablets: Results from all subjects following dosing with placebo tablets
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
percentage of time with pH below pH 4 | 5.14 [-0.27 to 10.56] | 14.94 [9.52 to 20.35]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -9.79, 95% CI 2-sided [-14.85 to -4.74]

2. Secondary Outcome: Percentage of Time During the 4-hour Post-dosing Period With pH Below pH 5
Description: Percentage of time during the 4-hour post-dosing period with pH below pH 5 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time with pH below pH 5
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
percentage of time with pH below pH 5 | 10.40 [3.40 to 17.40] | 26.16 [19.16 to 33.16]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -15.76, 95% CI 2-sided [-22.82 to -8.71]

3. Secondary Outcome: Number of Occasions During the 4-hour Post-dosing Period When pH Falls Below pH 4
Description: Number of occasions during the 4-hour post-dosing period when pH falls below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of occasions pH fell below 4
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
Number of occasions pH fell below 4 | 11.5 [3.4 to 19.6] | 30.9 [22.8 to 39.1]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Median Difference (Final Values) = -19.4, 95% CI 2-sided [-29.6 to -9.2]

4. Secondary Outcome: Number of Occasions During the 4-hour Post-dosing Period When pH Falls Below pH 5
Description: Number of occasions during the 4-hour post-dosing period when pH falls below pH 5 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of occasions pH fell below 5
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
Number of occasions pH fell below 5 | 17.3 [9.5 to 25.1] | 33.6 [25.8 to 41.4]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0019, Mixed Models Analysis; Mean Difference (Final Values) = -16.3, 95% CI 2-sided [-26.2 to -6.4]

5. Secondary Outcome: Number of Reflux Episodes During the 4-hour Post-dosing Period With pH Below pH 4 for at Least 5 Minutes
Description: Number of reflux episodes during the 4-hour post-dosing period with pH below pH 4 for at least 5 minutes for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of reflux episodes
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
Number of reflux episodes | 0.6 [-0.1 to 1.3] | 1.4 [0.7 to 2.1]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0290, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.6 to -0.1]

6. Secondary Outcome: Percentage of Time During the First Hour Post-dosing With pH Below pH 4
Description: Percentage of time during the first hour post-dosing with pH below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 1 hour post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time with pH below pH 4
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
percentage of time with pH below pH 4 | 2.00 [-3.43 to 7.44] | 16.41 [10.98 to 21.84]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -14.40, 95% CI 2-sided [-20.57 to -8.23]

7. Secondary Outcome: Percentage of Time During the First Hour Post-dosing With pH Below pH 5
Description: Percentage of time during the first hour post-dosing with pH below pH 5 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 1 hour post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time with pH below pH 5
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
percentage of time with pH below pH 5 | 4.23 [-2.82 to 11.29] | 27.60 [20.55 to 34.65]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -23.37, 95% CI 2-sided [-31.55 to -15.19]

8. Secondary Outcome: Number of Occasions During the First Hour Post-dosing When pH Falls Below pH 4
Description: Number of occasions during the first hour post-dosing when pH falls below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 1 hour post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of occasions pH fell below 4
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
Number of occasions pH fell below 4 | 1.7 [-0.6 to 4.0] | 9.1 [6.7 to 11.4]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-10.0 to -4.6]

9. Secondary Outcome: Number of Occasions During the First Hour Post-dosing When pH Falls Below pH 5
Description: Number of occasions during the first hour post-dosing when pH falls below pH 5 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 1 hour post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of occasions pH fell below 5
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
Number of occasions pH fell below 5 | 3.1 [0.8 to 5.4] | 9.5 [7.2 to 11.8]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-9.4 to -3.3]

10. Secondary Outcome: The Longest Reflux Time During the 4-hour Post-dosing Period (i.e. the Longest Period With pH Below pH 4)
Description: The longest reflux time during the 4-hour post-dosing period (i.e. the longest period with pH below pH 4) for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
minutes | 3.3 [-1.3 to 7.9] | 9.6 [5.1 to 14.2]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0075, Mixed Models Analysis; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-10.9 to -1.8]

11. Secondary Outcome: The DeMeester Scores During the 4-hour Post-dosing Period
Description: The DeMeester scores during the 4-hour post-dosing period for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets.
  The DeMeester score is a composite score of the acid exposure during a prolonged ambulatory pH monitoring. The parameters that constitute the score are number of reflux episodes, number of episodes longer than 5 minutes, longest reflux duration, total percentage of monitoring time with pH below 4, and the percentage of time with pH below 4 in an upright position and supine position, respectively. The DeMeester score is the sum of the scores calculated for each of the 6 parameters. A score more than 14.7 is considered abnormal acid reflux, scores between 14.7 and 100 are regarded as mild-to-moderate GERD, and a score greater than 100 is regarded as severe GERD.
Time Frame: 0 to 4 hours post-dose
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Placebo Tablets
Number analyzed (Participants) | 44 | 44
score on a scale | 14.842 [2.125 to 27.560] | 38.987 [26.270 to 51.704]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Placebo Tablets; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -24.145, 95% CI 2-sided [-37.432 to -10.858]

ADVERSE EVENTS:
Time Frame: Up to 19 days, from the time informed consent was provided until the Day 7 (+/- 2 days) visit
Description: In both reported AEs, blood samples, from which the TEAEs of "White blood cell count decreased" were identified, were taken 1 week after administration of 4 placebo tablets followed by 7 days of Sodium Alginate Double Action Chewable Tablets (2 tablets 4times daily), and ~4 hours after administration of 4 Sodium Alginate Double Action Chewable Tablets. It was not possible to definitely attribute these AEs to one or other of the interventions, so AEs are reported by group, not by intervention.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=22) | Group B (N=23)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-06-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT01872897/Prot_000.pdf
  • Statistical Analysis Plan (2014-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT01872897/SAP_001.pdf